CLINICAL TRIAL: NCT00734669
Title: Risk of Hypoglycemia in Type 2 Diabetes - Effects of Glibenclamide and Exercise on Cardiovascular, Hormonal, and Metabolic Parameters
Brief Title: Risk of Hypoglycemia in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Thomas Linn, Univ.-Prof. Dr. med., University of Giessen
Other Study IDs: EC 84/08
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypoglycemia | interventions — Glyburide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Type 2 diabetic patients on glibenclamide at individual dosage up to 7 mg/day for more than one year prone to hypoglycemic events
  Interventions: Drug: Glibenclamide

INTERVENTIONS:
Drug: Glibenclamide — Taking a single dose of 3.5 mg glibenclamide

SUMMARY:
The aim of this study is to establish the risk and frequency of non-symptomatic hypoglycemia in type 2 diabetes under previous therapy with glibenclamide. Participants will be monitored via a continuous glucose monitoring system in a standardized clinical setting during day and night time, implementing meals and exercise of moderate intensity performed in the postprandial state.

DETAILED DESCRIPTION:
The day-to-day change of blood glucose is associated with the frequency of vascular complications and the quality of life of diabetic patients. In this study the frequency of hypoglycemic events in combination with postprandial hyperglycemia in type 2 diabetic patients on oral insulinotropic therapy will be observed. Using more sophisticated technology than before the probability of type 2 diabetic patients on glibenclamide to experience hypoglycemic episodes will be registered. Hypoglycemia is prone to cardiovascular complications in type 2 diabetic patients due to concomitant dysregulation of blood flow. With standardized test meals followed by exercise in a clinical setting hormonal counterregulation and cardiovascular parameters associated with hypoglycemia will be identified. The acute effect of different conditions of exercise and a single dose of either glibenclamide or placebo will be followed each day during the total three-day observation period. Thus we will evaluate the frequency of and the risk factors associated with hypoglycemia and meal-related hyperglycemia in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on glibenclamide with or without
* Glycated hemoglobin ≤ 7.5%
* Stable dosage for three weeks

Exclusion Criteria:

* HbA1c > 7.5%
* Fasting C-peptide below normal
* Concurrent infectious disease
* Pregnancy
* Malignant disease
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic events | 3 days

SECONDARY OUTCOMES:
Secretion of hormones increasing blood glucose, effect of exercise on hypoglycemic events, postprandial glucose excursions, heart rate and forearm blood flow at hypoglycemia | 3 days

IPD SHARING:
Plan to Share IPD: No